CLINICAL TRIAL: NCT04892940
Title: Use of Virtual Reality to Reduce Morphine Consumption in Adolescents Undergoing Scoliosis Surgery: a Prospective Randomized Open-label Study. Virtual Reality for Analgesia in Spine Surgery
Brief Title: Use of Virtual Reality to Reduce Morphine Consumption in Adolescents Undergoing Scoliosis Surgery
Acronym: ViRAgeSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/20/0447
Record Dates: First submitted 2021-04-08; First posted 2021-05-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Scoliosis
Keywords: Virtual reality; Scoliosis surgery; Adolescents; Pain management
MeSH Terms: conditions — Scoliosis; Agnosia | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality group (Experimental): Adolescents aged 13 to 18 years who have undergone scoliosis surgery
  Interventions: Device: Virtual Reality (VR) technique; Drug: Analgesic protocol
- Control group (Active Comparator): Adolescents aged 13 to 18 years who have undergone scoliosis surgery
  Interventions: Drug: Analgesic protocol

INTERVENTIONS:
Device: Virtual Reality (VR) technique — The "PICO G2 4k" helmet from the Chinese manufacturer Pico which is an autonomous virtual reality helmet will be used.
  The sessions proposed last 20 minutes with a "child pain" protocol. The teenager will be able to choose his universe (forest, beach, mountain, aquatic, space), the voice that accompanies him (man, woman, none), the sound environment of music therapy (6 to choose from).
  Each patient in the experimental group benefits from a virtual reality program including two daily sessions during their stay in the continuing care unit from the first post-operative day until the third post-operative day. Each session is proposed by a nurse anesthetist from the pain team and trained in the proper use of the equipment.This virtual reality program will be added to the standard analgesic protocol for the experimental group.
  Arms: Virtual Reality group
Drug: Analgesic protocol — Patients randomized in the "control" group receive the usual analgesic protocol of the department postoperatively.

SUMMARY:
The objective is to evaluate the effect of the association of virtual reality sessions with usual management on the cumulative consumption of morphine equivalent post-operatively in adolescents aged 13 to 18 years who have undergone scoliosis surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 13 and 18 years old, i.e. the age to use a virtual reality helmet according to the manufacturer's recommendations.
* Patient with an indication for idiopathic scoliosis surgery.
* Free, informed and signed consent by patients (or parents/parental guardians) and the investigator (no later than the day of inclusion and prior to any review required by the research)

Exclusion Criteria:

* Patient undergoing surgery for neurological scoliosis.
* Impossibility to use the VR helmet (blindness, eye infection, helmet wound, epilepsy, psychiatric or cognitive disorder incompatible with VR).
* History of adverse effects while wearing an VR helmet (nausea, vomiting, headache, visual disturbances)
* Patient with a contraindication to the use of morphinics
* Patient whose both parents benefit from a legal protection measure (guardianship, curatorship, safeguard of justice)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Cumulative amount of morphine (mg) consumed for each participant. | From day 1 to day 3 postoperatively

SECONDARY OUTCOMES:
Intensity of pain assessed on a scale of 1 to 10. | At day 3 postoperatively
  The patient will assess his pain on a scale ranging from 1 to 10, 1 being a very low pain to 10 very strong pain.
Maximum level of pain assessed on a scale of 1 to 10 | From day 1 to day 6 postoperatively
  The patient will assess his pain on a scale ranging from 1 to 10, 1 being a very low pain to 10 very strong pain.
Morphine-related side effects | Between day 1 and day 3 postoperatively
  Number and nature of morphine-related side effects
Treatment prescribed to combat the side effects of morphine | Between day 1 and day 3 postoperatively
  Nature of treatment
Dose of treatment prescribed to combat the side effects of morphine | Between day 1 and day 3 postoperatively
  Dose in mg
Duration of treatment prescribed to combat the side effects of morphine | Between day 1 and day 3 postoperatively
  Number of days
daily dose of morphine | From day 1 to day 6 postoperatively
  daily dose of morphine equivalent in milligrams (mg) then related to the weight in milligrams per kilogram (mg/kg)
Cost-effectiveness ratio | From day 1 to day 6 postoperatively
  Calculated by taking into account the costs collected from the point of view of health insurance and the number of patients having avoided side effects at 6 days
Side effects related to the use of the virtual reality | From day 1 to day 3 postoperatively
  Number of side effects
Number of drug treatments as well as the purchase price of RV from a hospital perspective | From day 1 to day 6 postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Servane LE GOAS UGUEN, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No